## Study Title: Building Engagement using Financial Incentives Trial – Colorectal cancer screening (BENEFIT-C)

**NCT Number** 

NCT06124131

Statistical Analysis Plan Date: 3/11/2024

Version Date: 3/11/2024 Version Number: 4.0

Page 1 of 4

**BENEFIT-C Statistical Analysis Plan.** Analyses for the primary outcome will test the betweengroup difference in the proportion of participants who completed a colorectal cancer screening at 2-month follow-up. Secondary outcomes will test between-group differences in the proportion of participants completing a flu shot, COVID-19 shot, any of the three services, and all three services at 2-month follow-up. Analyses will use a chi-squared test of independence or a Fisher's exact test, as appropriate based on achieved cell sizes. We will also test for statistically significant betweengroup differences in baseline characteristics, and if necessary, adjust for them in a follow-up sensitivity analysis using multivariable logistic regression.